CLINICAL TRIAL: NCT06847750
Title: Elastography Ultrasound in Localized Scleroderma (Morphea): a Prospective, Longitudinal, Multicentric Pilot Study
Brief Title: Elastography Ultrasound in Localized Scleroderma (Morphea) Study
Status: Enrolling by invitation | Type: Observational
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Childhood Arthritis and Rheumatology Research Alliance (Other); Joseph Sanzari Children's Hospital (Unknown); University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Andrea Doria, Professor, Vice-Chair of Radiology (Clinical Practice Improvement), Department of Medical Imaging, University of Toronto Radiologist, Senior Scientist, Research Director, Department of Diagnostic Imaging, The Hospital for Sick Children
Other Study IDs: 1000078198
Record Dates: First submitted 2024-12-16; First posted 2025-02-26 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Scleroderma
Keywords: Elastography ultrasound; Scleroderma; Quality of Life; Pediatric
MeSH Terms: conditions — Scleroderma, Diffuse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Elastography group: Boys and girls 0-18 years of age at the time of disease onset with a new or existing diagnosis of localized scleroderma will have a physical examination and elastogrpahy ultrasound at specific timepoints, based on the timeframe for clinical visits. A questionnaire will be administered by the time of each study visit.
  Interventions: Diagnostic Test: Elastography Ultrasound; Other: The Localized Scleroderma Quality of Life Instrument (LoSQI )

INTERVENTIONS:
Diagnostic Test: Elastography Ultrasound — The US imaging protocol will include three parts: (i) gray-scale; (ii) color Doppler, and (iii) Shear-wave elastography (SWE)
Other: The Localized Scleroderma Quality of Life Instrument (LoSQI ) — The questionnaire is a validated disease-specific patient-reported outcome measure that covers different domains (skin sensations, physical functioning, body image and social support, designed for children and adolescents with localized scleroderma

SUMMARY:
Localized scleroderma (LS) is a skin disease that can cause complications such as disfigurement and limitation of mobility. Treatment for LS should be initiated early in the disease, as late-stage scleroderma does not respond well to treatment. Objective tools for diagnosis and follow-up of treatment for LS are not available clinically and are urgently needed. A new non-invasive ultrasound technique called "elastography" measures stiffness of tissues and holds potential for providing objective measures for follow-up of treatment of LS in children and adolescents. The team plans to conduct a multicenter study in North America to determine whether elastography ultrasound can show changes in skin stiffness for a period of 9 to 12 months after initiation of treatment for LS. This novel technology may add information to the existing imperfect clinical tools, thus improving the way therapy is offered to patients with LS.

ELIGIBILITY:
Inclusion Criteria:

* Boys and girls 0-18 years of age at the time of disease onset with a new or existing diagnosis of localized scleroderma (LS) confirmed by a pediatric rheumatologist or dermatologist.
* Presents with one active or inactive lesion, using the contralateral site for comparison at each visit, as long as the same lesion is evaluated at each time point. OR Presents with more than one lesion as far as both lesions are active or inactive.
* Able to cooperate with clinical and US evaluation, and the parent or guardian is able to fill out interim patient history form.

Exclusion Criteria:

* Patients with other co-morbidities (e.g. systemic sclerosis, juvenile idiopathic arthritis, other systemic diseases).
* Patients who present with one active and one inactive lesion.
* Patients with lesions located in the face or head.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with diagnosis of LS
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-03-10 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Skin stiffness | Baseline, 3-6m and 9-12m
  Skin stiffness will be assessed using Elastography (SWE) Ultrasound, a sonographic technique that uses mechanical waves to assess tissue elasticity and display it in a quantitative manner. The stiffness of the tissue is directly proportional to its shear wave velocity. SWE will measure interval changes of skin stiffness during treatment at the target lesion and the unaffected contralateral site.

SECONDARY OUTCOMES:
Lesion activity responsiveness | Baseline, 3-6m and 9-12m
  The LoSCAT (Localized Sclerodema Cutaneous Assessment Tool scores) assesses 18 cutaneous anatomic sites, capturing both disease activity (mLoSSI - Modified Localized Skin Severity Index) and disease damage (LoSDI - Localized Scleroderma Damage Index). Scores for each site are based on the most severe score for each parameter ranging from 0 to 3. A higher score represents a worse outcome.
Echogenicity scores for dermis and hypodermis | Baseline, 3-6m and 9-12m
  Standard ultrasound protocol. Identifying sonographic changes in the involved body site will be accomplished by comparing both echogenicity and color Doppler signal to a corresponding normal site. The score is determined by summing the absolute value of the individual parameters, with a range from 0 to 15 (maximum echogenicity score of 6, maximum vascularity score of 9). A higher score represents a worse outcome.
Vascularity scores for dermis and hypodermis | Baseline, 3-6m and 9-12m
  Doppler Ultrasound protocol. Identifying sonographic changes in the involved body site will be accomplished by comparing both echogenicity and color Doppler signal to a corresponding normal site. The score is determined by summing the absolute value of the individual parameters, with a range from 0 to 15 (maximum echogenicity score of 6, maximum vascularity score of 9). A higher score represents a worse outcome.
Quality of Life | Baseline, 3-6m and 9-12m
  Completiom of the LoSQI (Localized Scleroderma Quality of Life Instrument), a self-reported disease-specific questionnaire to assess the quality of life of patients (children, adolescents and young adults) with localized scleroderma. It consists of 21 items across three theoretical domains: (1) skin sensations, (2) physical functioning and musculoskeletal sequelae, and (3) body image and social support. Scores are based on the most severe score for each parameter ranging from 0 to 3.
  The questionnaire includes questions that comprise the Pain & Physical Functioning subscale, and the Body Image & Social Support subscale. Scores are summoned and converted to a scale, ranging from 41.3 to 71.6 and 43.58 to 68.42, respectively.
  A higher score represents a worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: CARRA is a registered non-profit organization. Its mission is to conduct collaborative research to prevent, treat and cure pediatric rheumatic diseases. — https://carragroup.org/grant/elastography-ultrasound-in-localized-scleroderma-morphea-a-prospective-longitudinal-multicentric-pilot-study-2/